CLINICAL TRIAL: NCT03752593
Title: The Incidence of Difficult Intubation in Obese Versus Non-obese Patients
Status: Completed | Type: Observational
Sponsor: King Hamad University Hospital, Bahrain (Other)
Responsible Party: Principal Investigator, Dr. Jaffar Albareeq, Director of Research, King Hamad University Hospital, Bahrain
Other Study IDs: KHUH/Anesthesia
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Obese: Patients with a BMI of greater than 30 who are presenting to the hospital for any surgical procedure requiring general anesthesia
  Interventions: Other: ET Tube
- Non-Obese: Patients with a BMI of less than 30 who are presenting to the hospital for any surgical procedure requiring general anesthesia
  Interventions: Other: ET Tube

INTERVENTIONS:
Other: ET Tube — Patients with a BMI of greater than 30 or less than who are presenting to the hospital for any surgical procedure requiring general anesthesia

SUMMARY:
The aim of our study is to identify the incidence of difficult endotracheal intubation in patients with normal BMI undergoing surgery under general anaesthesia in our hospital and compare it to that of obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* BMI< 30 for Normal BMI group
* BMI > 30 for Obese group

Exclusion Criteria:

* Known previous difficult airway
* Pediatric patients.
* Emergency patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heterogeneous group representing the general population of Muharraq
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Assessment of difficulty in airway management | two years
  Assessment of Cormack Lehanne grading (intubation difficulty scale) IDS.

CONTACTS AND LOCATIONS:
Locations (1):
- King Hamad University Hospital, Al Muharraq, Bahrain

REFERENCES:
- [Background] Murphy C, Wong DT. Airway management and oxygenation in obese patients. Can J Anaesth. 2013 Sep;60(9):929-45. doi: 10.1007/s12630-013-9991-x. Epub 2013 Jul 9. PMID 23836064
- [Background] Lundstrom LH. Detection of risk factors for difficult tracheal intubation. Dan Med J. 2012 Apr;59(4):B4431. PMID 22459727
- [Background] Shiga T, Wajima Z, Inoue T, Sakamoto A. Predicting difficult intubation in apparently normal patients: a meta-analysis of bedside screening test performance. Anesthesiology. 2005 Aug;103(2):429-37. doi: 10.1097/00000542-200508000-00027. PMID 16052126
- [Background] Lavi R, Segal D, Ziser A. Predicting difficult airways using the intubation difficulty scale: a study comparing obese and non-obese patients. J Clin Anesth. 2009 Jun;21(4):264-7. doi: 10.1016/j.jclinane.2008.08.021. Epub 2009 Jun 6. PMID 19502026
- [Background] Kim WH, Ahn HJ, Lee CJ, Shin BS, Ko JS, Choi SJ, Ryu SA. Neck circumference to thyromental distance ratio: a new predictor of difficult intubation in obese patients. Br J Anaesth. 2011 May;106(5):743-8. doi: 10.1093/bja/aer024. Epub 2011 Feb 24. PMID 21354999
- [Background] De Jong A, Molinari N, Pouzeratte Y, Verzilli D, Chanques G, Jung B, Futier E, Perrigault PF, Colson P, Capdevila X, Jaber S. Difficult intubation in obese patients: incidence, risk factors, and complications in the operating theatre and in intensive care units. Br J Anaesth. 2015 Feb;114(2):297-306. doi: 10.1093/bja/aeu373. Epub 2014 Nov 27. PMID 25431308
- [Background] Juvin P, Lavaut E, Dupont H, Lefevre P, Demetriou M, Dumoulin JL, Desmonts JM. Difficult tracheal intubation is more common in obese than in lean patients. Anesth Analg. 2003 Aug;97(2):595-600. doi: 10.1213/01.ANE.0000072547.75928.B0. PMID 12873960
- [Background] Hashim MM, Ismail MA, Esmat AM, Adeel S. Difficult tracheal intubation in bariatric surgery patients, a myth or reality? Br J Anaesth. 2016 Apr;116(4):557-8. doi: 10.1093/bja/aew039. No abstract available. PMID 26994235
- [Background] Karkouti K, Rose DK, Wigglesworth D, Cohen MM. Predicting difficult intubation: a multivariable analysis. Can J Anaesth. 2000 Aug;47(8):730-9. doi: 10.1007/BF03019474. PMID 10958088
- [Background] Brodsky JB, Lemmens HJ, Brock-Utne JG, Vierra M, Saidman LJ. Morbid obesity and tracheal intubation. Anesth Analg. 2002 Mar;94(3):732-6; table of contents. doi: 10.1097/00000539-200203000-00047. PMID 11867407
- [Background] Bond A. Obesity and difficult intubation. Anaesth Intensive Care. 1993 Dec;21(6):828-30. doi: 10.1177/0310057X9302100614. No abstract available. PMID 8122742
- [Background] Benumof JL. Management of the difficult adult airway. With special emphasis on awake tracheal intubation. Anesthesiology. 1991 Dec;75(6):1087-110. doi: 10.1097/00000542-199112000-00021. PMID 1824555
- [Background] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827